CLINICAL TRIAL: NCT07328009
Title: The HCC-SIGHT: A Therapy Platform Trial for Hepatocellular Carcinoma Guided by Stratification Imaging and Genetic Horizon Testing
Brief Title: A Platform Trial for Personalized and Adaptive Therapies in Hepatocellular Carcinoma
Acronym: HCC-SIGHT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Peng Wang, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC-SIGHT
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Hepato Cellular Carcinoma (HCC)
MeSH Terms: interventions — lenvatinib; regorafenib; ursodoxicoltaurine; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- TKI (Control Therapy) (Active Comparator): Lenvatinib OR Regorafenib
  Interventions: Drug: Lenvatinib; Drug: Regorafenib (BAY 73-4506)
- Tislelizumab+TKI (Experimental): Tislelizumab+TKI
  Interventions: Drug: Tislelizumab+TKI
- HAIC+TKI (Experimental): HAIC (Hepatic Arterial Infusion Chemotherapy)+TKI
  Interventions: Drug: HAIC+TKI
- HAIC + Tislelizumab+TKI (Experimental): HAIC + Tislelizumab+TKI
  Interventions: Drug: HAIC + Tislelizumab+TKI
- QL1706+TKI (Experimental): QL1706 (iparomlimab/tuvonralimab)+TKI
  Interventions: Drug: QL1706+TKI
- HAIC + QL1706+TKI (Experimental): HAIC + QL1706+TKI
  Interventions: Drug: HAIC + QL1706+TKI
- TUDCA + Camrelizumab+TKI (Experimental): TUDCA + Camrelizumab+TKI
  Interventions: Drug: TUDCA + Camrelizumab+TKI
- XELOX + Tislelizumab+TKI (Experimental): XELOX (chemotherapy) + Tislelizumab+TKI
  Interventions: Drug: XELOX + Tislelizumab+TKI
- XELOX + QL1706+TKI (Experimental): XELOX (chemotherapy) + Tislelizumab+TKI
  Interventions: Drug: XELOX + QL1706+TKI

INTERVENTIONS:
Drug: Lenvatinib — 12 mg orally daily for body weight ≥ 60 kg; 8 mg orally daily for body weight < 60 kg.
  Arms: TKI (Control Therapy)
Drug: Regorafenib (BAY 73-4506) — 160 mg orally once daily on Days 1-21 of a 28-day cycle.
  Arms: TKI (Control Therapy)
Drug: Tislelizumab+TKI — Tislelizumab:200 mg administered intravenously (IV) on Day 1 of each 21-day cycle.
  Lenvatinib：8 mg orally daily；OR Regorafenib：80 mg orally once daily on Days 1-21 of a 28-day cycle.
  Arms: Tislelizumab+TKI
Drug: HAIC+TKI — FOLFOX Regimen: Administered via the hepatic artery. Oxaliplatin: 85 mg/m² IV infusion from Hour 0-2 on Day 1. Leucovorin: 400 mg/m² IV infusion from Hour 2-3 on Day 1. Fluorouracil: 400 mg/m² IV bolus at Hour 3 on Day 1, followed by 2400 mg/m² as a continuous IV infusion over 24 hours.
  HAIC was repeated every 3 weeks for up to 4 cycles. Lenvatinib：8 mg orally daily；OR Regorafenib：80 mg orally once daily on Days 1-21 of a 28-day cycle.
  Arms: HAIC+TKI
Drug: HAIC + Tislelizumab+TKI — FOLFOX Regimen: Administered via the hepatic artery. Oxaliplatin: 85 mg/m² IV infusion from Hour 0-2 on Day 1. Leucovorin: 400 mg/m² IV infusion from Hour 2-3 on Day 1. Fluorouracil: 400 mg/m² IV bolus at Hour 3 on Day 1, followed by 2400 mg/m² as a continuous IV infusion over 24 hours.HAIC was repeated every 3 weeks for up to 4 cycles.
  Tislelizumab: 200 mg IV on Day 1 of each 21-day cycle. Lenvatinib：8 mg orally daily；OR Regorafenib：80 mg orally once daily on Days 1-21 of a 28-day cycle.
  Arms: HAIC + Tislelizumab+TKI
Drug: QL1706+TKI — QL1706:7.5 mg/kg IV on Day 1 of each 21-day cycle. Lenvatinib：8 mg orally daily；OR Regorafenib：80 mg orally once daily on Days 1-21 of a 28-day cycle.
  Arms: QL1706+TKI
Drug: HAIC + QL1706+TKI — FOLFOX Regimen: Administered via the hepatic artery. Oxaliplatin: 85 mg/m² IV infusion from Hour 0-2 on Day 1. Leucovorin: 400 mg/m² IV infusion from Hour 2-3 on Day 1. Fluorouracil: 400 mg/m² IV bolus at Hour 3 on Day 1, followed by 2400 mg/m² as a continuous IV infusion over 24 hours. HAIC was repeated every 3 weeks for up to 4 cycles.
  QL1706: 7.5 mg/kg IV on Day 1 of each 21-day cycle. Lenvatinib：8 mg orally daily；OR Regorafenib：80 mg orally once daily on Days 1-21 of a 28-day cycle.
  Arms: HAIC + QL1706+TKI
Drug: TUDCA + Camrelizumab+TKI — Tauroursodeoxycholic Acid (TUDCA): 250 mg orally twice daily. Camrelizumab: 200 mg IV on Day 1 of each 14-day cycle. Lenvatinib：8 mg orally daily；OR Regorafenib：80 mg orally once daily on Days 1-21 of a 28-day cycle.
  Arms: TUDCA + Camrelizumab+TKI
Drug: XELOX + QL1706+TKI — Oxaliplatin, 85 mg/m² IV infusion on Day 1 every 3 weeks; Capecitabine, 1000 mg/m2, orally twice daily on days 1 to 14 every 3 weeks. XELOX was repeated every 3 weeks for up to 4 cycles. QL1706: 7.5 mg/kg IV on Day 1 of each 21-day cycle. Lenvatinib：8 mg orally daily；OR Regorafenib：80 mg orally once daily on Days 1-21 of a 28-day cycle.
  Arms: XELOX + QL1706+TKI
Drug: XELOX + Tislelizumab+TKI — Oxaliplatin, 85 mg/m² IV infusion on Day 1 every 3 weeks; Capecitabine, 1000 mg/m2, orally twice daily on days 1 to 14 every 3 weeks.
  XELOX was repeated every 3 weeks for up to 4 cycles. Tislelizumab: 200 mg IV on Day 1 of each 21-day cycle. Lenvatinib：8 mg orally daily；OR Regorafenib：80 mg orally once daily on Days 1-21 of a 28-day cycle.
  Arms: XELOX + Tislelizumab+TKI

SUMMARY:
This is a phase II, multi-arm, Bayesian adaptive platform trial designed to efficiently evaluate novel therapies for advanced hepatocellular carcinoma (HCC) after first-line treatment failure. The study aims to rapidly identify the most effective investigational regimens and discover predictive biomarker signatures (from tumor tissue, blood, and imaging) to guide personalized second-line therapy.

DETAILED DESCRIPTION:
This open-label, adaptive platform trial addresses the lack of effective second-line therapies for advanced HCC. Multiple experimental regimens will be evaluated against a common control arm. The study employs a Bayesian adaptive design. Patient randomization probabilities will favor regimens showing better interim efficacy (primary endpoint: objective response rate). Underperforming regimens will be dropped, and new ones may be added over time. A key objective is to identify predictive biomarker signatures. Baseline and on-treatment biomarker assessments (including tumor molecular profiling, ctDNA, and quantitative imaging features) will be analyzed to define patient subsets most likely to respond to each therapy. Regimens with a high predictive probability of success will graduate for further development. Those with low probability of benefit will be discontinued. This design enables rapid, biomarker-informed therapy screening for second-line HCC.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Age ≥ 18 years at time of study entry.
* Locally advanced or metastatic and/or unresectable HCC with diagnosis confirmed by histology/ cytology or clinically by American Association for the Study of Liver Diseases (AASLD) criteria in cirrhotic patients.
* Patients who have previously received first-line therapy with anti-PD-1/PD-L1 combined with anti-VEGF antibodies, or anti-PD-1/PD-L1 combined with TKI, or anti-PD-1/PD-L1 combined with anti-CTLA-4 antibodies and experienced disease progression; or disease recurrence within 6 months after completion of neoadjuvant/adjuvant immunotherapy.
* At least one measurable (per RECIST v1.1) target lesion that has not been previously treated with local therapy or, if the target lesion is within the field of previous local therapy, has subsequently progressed in accordance with RECIST v1.1.
* Child-Pugh scores 5-7, performance status (PS) ≤ 2 (ECOG scale).
* Subjects with chronic HBV infection must have HBV DNA viral load < 100 IU/mL at screening. In addition, they must be on antiviral therapy per regional standard of care guidelines prior to initiation of study therapy.
* Life expectancy of at least 12 weeks.
* Adequate blood count, liver-enzymes, and renal function: absolute neutrophil count ≥ 1,500/L, platelets ≥60 x103/L; Total bilirubin ≤ 3x upper normal limit; Aspartate Aminotransferase (SGOT), Alanine aminotransferase (SGPT) ≤ 5 x upper normal limit (ULN); International normalized ratio (INR) ≤1.25; Albumin ≥ 31 g/dL; Serum Creatinine ≤ 1.5 x institutional ULN or creatinine clearance (CrCl) ≥ 30 mL/min (if using the Cockcroft-Gault formula)
* Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment, adherence to contraceptive measures, scheduled visits and examinations including follow up.

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
* Patients on a liver transplantation list or with advanced liver disease.
* History of cardiac disease, including clinically significant gastrointestinal bleeding within 4 weeks prior to start of study treatment
* Thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months Prior to the first dose of study drug with the exception of thrombosis of a segmental portal vein.
* Patients with second primary cancer, except adequately treated basal skin cancer or carcinoma in-situ of the cervix.
* Immunocompromised patients, e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Participation in another clinical study with an investigational product during the last 30 days before inclusion or 7 half-lifes of previously used trial medication, whichever is longer.
* Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study Treatment or interpretation of patient safety or study results, including but not limited to: a) history of interstitial lung disease b) Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) coinfection (i.e double infection) c) known acute or chronic pancreatitis d) active tuberculosis e) any other active infection (viral, fungal or bacterial) requiring systemic therapy f) history of allogeneic tissue/solid organ transplant g) diagnosis of immunodeficiency or patient is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of treatment. h) Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Exceptions: Subjects with vitiligo, hypothyroidism, diabetes mellitus type I or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with Hashimoto thyroiditis, hypothyroidism stable on hormone replacement or psoriasis not requiring treatment are not excluded from the study. i) Live vaccine within 30 days prior to the first dose of treatment or during study treatment. j) History or clinical evidence of Central Nervous System (CNS) metastases Exceptions are: Subjects who have completed local therapy and who meet both of the following criteria: I. are asymptomatic and II. have no requirement for steroids 6 weeks prior to start of treatment. Screening with CNS imaging (CT or MRI) is required only if clinically indicated or if the subject has a history of CNS.
* Medication that is known to interfere with any of the agents applied in the trial.
* Any other efficacious cancer treatment except protocol specified treatment at study start.
* Patient has received any other investigational product within 28 days of study entry.
* Female subjects who are pregnant, breast-feeding or male/female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year). [Acceptable methods of contraception are: implants, injectable contraceptives, combined oral contraceptives, intrauterine pessars (only hormonal devices), sexual abstinence or vasectomy of the partner]. Women of childbearing potential must have a negative pregnancy test (serum β-HCG) at screening.
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2029-01-15 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  ORR is defined as the percentage of participants who have a confirmed complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters). Responses are according to RECIST 1.1 as assessed by investigator.

SECONDARY OUTCOMES:
Disease control rate (DCR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  DCR is defined as the proportion of patients with complete response (CR), partial response (PR) and stable disease (SD).
Duration of Response (DOR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  DOR is defined as the time from first documented complete or partial response until disease progression, death from any cause, or censoring at date of last tumor assessment.
Time to Response (TTR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1. | max 24 months
  TTR is defined as the time from the start of treatment until the first objective observation of a response (either partial response, PR, or complete response, CR), provided that the response is subsequently confirmed.
Progression Free Survival (PFS) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1. | max 24 months
  PFS is defined as the time from study treatment to disease progression or all-cause death as assessed by the investigator (whichever occurs first).
Overall survival (OS) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1. | max 42 months
  OS is defined as the time from study treatment to the date of death of the subject, regardless of the cause of death.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | max 42 months
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experience at least one AE will be reported.
Translational study. | max 42 months
  To identify predictive biomarker signatures. Baseline and on-treatment biomarker assessments (including tumor molecular profiling, ctDNA, and quantitative imaging features) will be analyzed to define patient subsets most likely to respond to each therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No